CLINICAL TRIAL: NCT06117280
Title: Effect of Different Dosages of Paraxanthine, the Major Caffeine Metabolite, on Energy and Focus: A Randomized, Double-Blind, Placebo-Controlled, Crossover Trial
Brief Title: Effect of Different Dosages of Paraxanthine, the Major Caffeine Metabolite, on Energy and Focus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iovate Health Sciences International Inc (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 20329
Record Dates: First submitted 2023-10-25; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Energy; Focus; Caffeine Withdrawal
MeSH Terms: interventions — 1,7-dimethylxanthine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention (Dose One) (Experimental): In this crossover trial, all participants will test both active comparators and the placebo comparator.
  Interventions: Other: Paraxanthine 200 mg
- Intervention (Dose Two) (Experimental): In this crossover trial, all participants will test both active comparators and the placebo comparator.
  Interventions: Other: Paraxanthine 300 mg
- Placebo (Placebo Comparator): In this crossover trial, all participants will test both active comparators and the placebo comparator.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Paraxanthine 200 mg — For the three-day test cycle, participants will take one capsule per day amounting to 200mg of paraxanthine.
  Arms: Intervention (Dose One)
Other: Paraxanthine 300 mg — For the three-day test cycle, participants will take one capsule per day amounting to 300mg of paraxanthine.
  Arms: Intervention (Dose Two)
Other: Placebo — The placebo will contain resistant dextrin. For the three-day test cycle, participants will take one capsule per day amounting to 300mg of resistant dextrin.
  Arms: Placebo

SUMMARY:
Research has shown that acute ingestion of Paraxanthine (1,7-dimethylxanthine, PXN) can enhance various markers of focus, including memory, reaction time, and attention in healthy adults. To assess these effects, this placebo-controlled crossover trial will compare the effects of 200 and 300mg of PXN to a placebo control. Participants will abstain from caffeine for 3 days, before taking the first test/placebo product for 3 consecutive days. Participants will complete questionnaires at 30, 60, 90, and 120 minutes after ingestion on Day 1 and Day 3 of ingestion. Participants will have a 3-day washout period before trialing the next test product/placebo.

DETAILED DESCRIPTION:
Following enrollment to the study, participants will abstain from any products containing caffeine, for 3 days.

On the night of the 3rd day of caffeine abstinence, participants will fast overnight (~10 hours) The morning after the fast, participants will complete the Day 1 baseline questionnaire.

Participants will then consume Test Product A and complete questionnaires 30, 60, 90, and 120 minutes after ingestion. Test Products should be consumed in a fasted state, and 1-hour post-ingestion participants will consume a standardized meal (See Section 6.3).

On Day 2, participants will consume Test Product A again but will not complete any questionnaires. The product should be consumed in a fasted state and participants will consume the standardized meal 60 minutes post-ingestion.

On Day 3, participants will consume Test Product A in a fasted state and will again consume the standardized meal 1-hour following ingestion of the product. Participants will complete questionnaires 30, 60, 90, and 120 minutes after ingestion. Participants will then have a 3-day washout period with no products consumed or questionnaires completed.

Following the washout period, the intervention cycle will be repeated with Test Product B and, subsequently, Test Product C.

The questionnaires will consist of study-specific surveys and a cognitive assessment battery.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-35
* Willing to abstain from caffeine-containing beverages and foods during the duration of the study
* Recreationally active; currently performing structured exercise (e.g., running, weightlifting, team-sport activity) at least 2 days per week for the previous 3 months

Exclusion Criteria:

* Body Mass Index: >29.9kg/m2
* Inability to adhere to protocol guidelines (e.g., caffeine, alcohol, tobacco)
* Regular tobacco use
* Illicit drug use (e.g., growth hormone, testosterone, etc.)
* A diagnosed medical condition under the care of a physician (e.g. type 2 diabetes) Inability to abstain from supplements (e.g. protein, creatine, HMB, BCAA, phosphatidic acid, etc.) at least three weeks before the trial
* Individuals on medications known to affect caffeine metabolism (e.g., corticosteroids, non-steroidal anti-inflammatories, or prescription-strength acne medications)
* Participants who are amenorrheic (females only)
* Inability to comply with the study protocol as judged by the investigators

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2023-07-18 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Changes in scores on a cognitive assessment "Double Trouble". [Time Frame: Baseline to Day 3 of each test cycle] | 18 days
  Participants will independently complete a cognitive assessment battery at home on their computer or tablet. "Double Trouble" is a 90-second timed test. Based on a classic Stroop test, Double Trouble measures selective attention, processing speed, and the brain's ability to focus on specific information when presented with conflicting and layered stimuli.
Changes in scores on a cognitive assessment "Feature Match". [Time Frame: Baseline to Day 3 of each test cycle] | 18 days
  Participants will independently complete a cognitive assessment battery at home on their computer or tablet. "Feature Match" is a 90-second timed test. Feature Match is a focus and processing task that requires surveying an increasingly difficult array of information and rapidly assessing the correct response while holding previously processed and detailed information in attention.
Changes in scores on a cognitive assessment "Grammatical Reasoning". [Time Frame: Baseline to Day 3 of each test cycle] | 18 days
  Participants will independently complete a cognitive assessment battery at home on their computer or tablet. "Grammatical Reasoning" is a 90-second timed test. Grammatical Reasoning is a deductive reasoning task that requires quickly interpreting phrases and making logical conclusions from understanding. Variation between text and shapes on screen requires holding key information in short-term memory to properly complete the task, leveraging the same parts of the brain that enable an individual to remain focused between varied stimuli.
Changes in scores on a cognitive assessment "Digit Span". [Time Frame: Baseline to Day 3 of each test cycle] | 18 days
  Participants will independently complete a cognitive assessment battery at home on their computer or tablet. "Digit Span is a 3-4 minute performance based test. Increasing in length after each successful attempt, Digit Span requires users to focus on displayed numbers, hold them in short-term memory, and repeat them back correctly, thereby showing cognitive flexibility and the brain's ability to perform memory and attention-related tasks without error.

SECONDARY OUTCOMES:
Occurence of the side effects of caffeine withdrawal. [Baseline to Endline] | 18 days
  Decrease in symptoms of caffeine withdrawal including jitters, fatigue, drowsiness, irritability, "brain fog", and low alertness. This will be reported via participant-reported questionnaires. Incidence and severity of side effects will be reported using a Likert scale (0-5 point scale) with 0=least severe and 5=most severe.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided